CLINICAL TRIAL: NCT00624975
Title: A Multi-site, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Immunogenicity of Trehalose-reformulated Peru-15 (Choleragarde)Vaccine Given Simultaneously With Measles Vaccine in Healthy Indian and Bangladeshi Infants
Brief Title: Safety and Immunogenicity of Peru-15 Vaccine When Given With Measles Vaccine in Healthy Indian and Bangladeshi Infants
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: one of site was not able to get an approval from the national regulatory authority.
Sponsor: International Vaccine Institute (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Christian Medical College, Vellore, India (Other); Avant Immunotherapeutics (Industry); Vaccine Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CHPR-01
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Cholera; Diarrhea; Vibrio Infections
MeSH Terms: conditions — Cholera; Diarrhea; Vibrio Infections | interventions — Peru 15

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccine (Experimental)
  Interventions: Biological: Peru-15 Vaccine
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Peru-15 Vaccine — up to 1 x 10^9 CFU of Peru-15 given in 5ml single dose vials with 20 ml buffer solution, given once
  Other Names: CholeraGarde
  Arms: Vaccine
Biological: Placebo — 25 mL of buffer solution (2.5 g sodium bicarbonate and 1.65 g ascorbic acid per 100mL potable water)
  Arms: Placebo

SUMMARY:
The purpose of this study is to confirm the safety and immunogenicity of Peru-15 vaccine in infants when given simultaneously with measles vaccine.

DETAILED DESCRIPTION:
Cholera is an important public health problem worldwide, remaining endemic in most of the developing world at the same time causing outbreaks in areas where lapses in sanitation occur. In 2005, 131 943 cholera cases and 2272 deaths were reported to the World Health Organization (WHO) with more countries reporting cholera outbreaks. Overall, this represents a 30% increase in the number of cases reported compared to 2004. The cholera case fatality rate during that year was 1.72%; however, recent outbreaks in West Africa resulted in case-fatality rates of as high as 12% [1, 2]. These figures are believed to be underestimates and that as much as 120 000 deaths due to cholera are estimated to occur each year [3]. Aside from this high mortality, cholera outbreaks cause economic and social disruptions.

The states of West Bengal in India together with neighboring Bangladesh have been considered by many as the "homeland of cholera". In India, 4695 cases of cholera were reported to the WHO [1] with states such as West Bengal, Maharashtra, Andra Pradesh, Tamil Nadu, Karnataka and Delhi long been reporting outbreaks [4]. Although no country-wide data is available from Bangladesh, a 4 - year surveillance in 4 different geographical areas in Bangladesh reveal that cholera is widely distributed even in an area with no reported outbreaks for 10 years [5]. Cholera in these 2 countries affects all age groups, with the youngest age group being the most affected. In Kolkata, children <5 years of age had a 30% higher risk of having cholera compared to older individuals [6] and in Bangladesh, 53% of 5670 cholera-infected patients in the 4-year surveillance were children <5 years of age [5]. Further analysis of a 3 year prospective surveillance of cholera in Kolkata shows that infants less than 2 years of age had a cholera incidence rate of 4.20 per 1000 person-years whereas the over-all rate in the study population was 1.41 per 1000 person-years (Data on file).

Provision of safe water and food, establishment of adequate sanitation, and implementation of personal and community hygiene constitute the main public health interventions against cholera. These measures cannot be fully implemented in the near future in most cholera-endemic areas. A safe, effective, and affordable vaccine would be a useful tool for cholera prevention and control.

Considerable progress has been made during the last decade in the development of new generation oral vaccines against cholera. These have already been licensed in some countries and are now being considered for wider public health application. The World Health Organization recently recommended that the newer generation cholera vaccines be considered in certain endemic and epidemic situations, but indicated that demonstration projects are needed to provide more information about the costs, feasibility, and impact of using these vaccines [7].

A killed oral cholera vaccine (Dukoral™) has long been available internationally, however its 2-dose schedule, the use of a buffer and the cost of the vaccine have impeded its use in public health settings. A live oral vaccine, CVD-103 HgR (Orochol™), although internationally licensed is currently not available in the market. This vaccine is only available for use in children older than 6 years old and adults. Despite the immunogenicity and efficacy in challenge studies in North American volunteers [8], in a field trial of this vaccine in an endemic area in Indonesia, no protective efficacy was detected during the period of observation [9].

A need exists for an improved cholera vaccine that is more thermostable and may be used in endemic countries in younger age groups. This new generation oral cholera vaccine must be administered in a single-dose regimen, be thermostable, confer high grade long-term protection and may be given to children below 2 years of age through mass immunization campaigns or through the expanded programme on immunization (EPI). In the Diseases of the Most Impoverished Programme (DOMI) of the IVI, Peru-15 was identified as the most promising of all the vaccine candidates. It is a live oral attenuated cholera vaccine derived from V. cholerae O1 El Tor Inaba strain that was first isolated in Peru in 1991 [10]. This has the advantage of being given in a single dose and of having the same biotype as the current pandemic strain (biotype El tor), unlike CVD-103 HgR which is a classical biotype. Peru-15 has been attenuated by several genetic modifications and deletions. By the deletion of the ctx A and the rtxA genes, it has been rendered unable to encode for cholera toxin subunit A and RTX toxin making it non-toxigenic and by insertion of the cholera toxin B gene to the recA gene, it enabled the strain to produce cholera toxin B. This insertion has inactivated the recA gene, and this together with the deletion of the attRS1 sequences, has decreased the ability of the strain to integrate exogenous DNA making it non-recombinational. Lastly, by the absence of the potentially inflammatory flagella it has been rendered non-motile [10, 11]. In addition, Phase I and II studies have been performed in North American volunteers where it was found to be safe and immunogenic [11-12]. Furthermore, the vaccine strain isolated from the stools of volunteers retained its non-motile characteristic. In a challenge study among North American volunteers, Peru-15 provided 100% protection against moderate and severe diarrhoea, and 93% against any diarrhoea [13].

This vaccine underwent phase I and II studies in a cholera-endemic area in Dhaka, Bangladesh in three age groups: adults aged 18 - 45 years, children aged 2 - 5 years and infants aged 9 - 23 months [14, 15]. In these studies, a 2 x108 CFU dose of the vaccine was shown to be safe and able to elicit vibriocidal responses among all age groups. 75% of adults, 84% of children aged 2-5 years and 70% of infants aged 9-23 months developed a 4-fold rise from baseline in their vibriocidal titres. Only 1 of 20 adults and 8 of 140 children who received vaccine excreted the vaccine strain up to 4 days after vaccination. Analysis of the strains isolated revealed that the strains remained unchanged in phenotypic and genotypic properties after passage in the stool.

To date, the vaccine has been tested on more than 400 volunteers. The freshly harvested product, tested on 23 volunteers and the frozen lyophilized preparation, tested on 381 volunteers were both shown to be safe and immunogenic in all age groups. The most frequently reported adverse events were gastrointestinal symptoms (diarrhea, nausea, abdominal cramping, gas, decreased appetite) and headache and in controlled studies were reported in similar frequencies in subjects who received Peru-15 and placebo. The optimal dose for healthy adult travelers was a single, oral dose of 1 x 108 CFU. The study in Bangladesh further confirmed that a 108 dose was safe and immunogenic in all age groups including infants among residents of a cholera endemic area.

Avant Immunotherapeutics Inc., manufacturers of Peru-15, are in the process of reformulating the vaccine with the long-term stabilizing ability of trehalose in order to make Peru-15 more thermostable at elevated temperatures, i.e. 2-8ºC. If this reformulation is proven as safe and at least as immunogenic as the previous version, then this will make vaccine storage easier and more easily deployable in field conditions in Africa, in refugee settings and in endemic countries in South Asia.

The International Vaccine Institute (IVI) through the Cholera Vaccine Initiative (CHOVI) together with Avant Immunotherapeutics Inc., manufacturers of the Peru-15 vaccine, have negotiated an agreement that allow clinical trials on this reformulated vaccine to be performed in 2 cholera-endemic countries - India and Bangladesh. This will eventually enable licensure and facilitate the international use of this vaccine by obtaining a WHO recommendation for its global use. This single dose vaccine may easily be used in endemic countries and deployed at times when outbreaks are likely to occur. Furthermore, this vaccine may potentially be used in infants and young children who have the highest risk of cholera, potentially being included as part of the EPI in endemic areas.

The previous formulations of the vaccine were shown to be safe and immunogenic in all age groups, including infants, in a cholera endemic area [12 - 15] and efficacious in preventing cholera diarrhea in healthy adult volunteers [13]. In view of this, the current dose of up to 109 of the current formulation will be directly tested among infants.Data regarding the safety and immunogenicity of the trehalose-reformulated Peru-15 vaccine among infants need to be confirmed in order to pave the way for the possible use of this vaccine in cholera-endemic areas where infants and children are most at risk. Furthermore, if this vaccine will be used in the context of the EPI to be given together with measles vaccine, it would be important to determine if immune interference exists between these 2 live attenuated vaccines.

ELIGIBILITY:
Inclusion Criteria:

Healthy male and female infants aged 9 - 12 months will be recruited from Vellore, India and Dhaka, Bangladesh.

All subjects must satisfy the following criteria at study entry:

1. Male or female infants aged 9 - 12 months whose parents or primary caretaker have given the written informed consent prior to study entry
2. Will comply with the requirements of the protocol (i.e. available for follow-up visits and specimen collection).
3. Healthy subjects as determined by:

   * Medical history
   * Physical examination
   * Clinical judgment of the investigator

Exclusion Criteria:

1. Parents or primary caregiver are unwilling or unable to give written informed consent to participate in the study
2. Ongoing serious chronic disease
3. Immunocompromising condition or therapy
4. Abdominal pain or cramps, loss of appetite, nausea, general ill-feeling or vomiting in the past 24 hours
5. Intake of any anti-diarrheal medicine in the past week
6. Acute disease one week prior to enrollment, with or without fever. Temperature ≥38ºC (oral) or axillary temperature ≥ 37.5ºC warrants deferral of the vaccination pending recovery of the subject
7. Receipt of antibiotics in the past 2 weeks
8. Receipt of live or killed enteric vaccine in the last 4 weeks
9. Diarrhea (3 or more loose stools within a 24-hour period) 6 weeks prior to enrollment
10. One or two episodes of diarrhea lasting for more than 2 weeks in the past 6 months
11. One or two episodes of abdominal pain lasting for more than 2 weeks in the past 6 months
12. Receipt of killed oral cholera vaccine
13. Have previously received a dose of a measles-containing vaccine (MCV)
14. Have previously presented with a disease potentially related to measles
15. Receipt of blood, blood products or a parenteral immunoglobulin preparation in the previous 3 months
16. History of anaphylaxis, any serious vaccine reaction, allergy to eggs, egg products or to any measles vaccine component
17. any condition which in the opinion of the investigator, might interfere with the evaluation of the study objectives

Ages: 9 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2008-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
proportion of subjects with the following adverse events: headache, vomiting, nausea, abdominal pain/cramps, gas, diarrhea, loss of appetite, myalgias, general ill feeling | 28 days
proportion of subjects exhibiting 4-fold or greater rises in titers of serum vibriocidal antibodies to serogroup O1 El Tor Inaba | relative to baseline, 1 week after dose
proportion of subjects who develop >150 mIU/ml measles IgG antibodies | 28 days after dose

SECONDARY OUTCOMES:
evaluate fecal excretion and genetic stability of the vaccine strain | 1,3,7,14 days after dosing
compare proportion of subjects given vaccine or placebo with any of the following adverse events: immediate events 30 minutes after dosing, serious adverse events throughout the trial | 30 minutes for adverse events, 28 days for serious adverse events
geometric mean serum vibriocidal, IgG anti-CTB and IgG anti-LPS (serogroup O1) antibody titers after vaccine or placebo | baseline and 1 week after dose

CONTACTS AND LOCATIONS:
Overall Officials: John Clemens, MD, Principal Investigator — International Vaccine Insititute
Locations (2):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh
- Christian Medical College, Vellore, India